CLINICAL TRIAL: NCT01135784
Title: Human CT: Efficacy & Safety of MIGRA-ZEN RELIEF PLUS:Herbal Supp:Extracts Juniper Willow Goldenrod Dandelion Meadowsweet Whole Grape In Rx of Chronic Migraine Headache. Randomized, Double-Blind, Placebo Cont. Study P.II (PoC Study)
Brief Title: Study of MIGRA-ZEN RELIEF PLUS In the Treatment of Chronic Migraine Headache
Acronym: RZN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RZN Nutraceuticals, Inc. (Industry)
Responsible Party: Mark Lubin, CEO & Chief Scientist, RZN Nutraceutricals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RZN 1
Record Dates: First submitted 2010-05-26; First posted 2010-06-03 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIGRA-ZEN RELIEF PLUS (Active Comparator): Active treatment
  Interventions: Dietary Supplement: MIGRA-ZEN RELIEF PLUS
- Placebo for Migra zen plus (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo for Migrazen relief plus

INTERVENTIONS:
Dietary Supplement: MIGRA-ZEN RELIEF PLUS — one 2-capsule dose per 24hrs for a total of 180 caps over 90 days
  Arms: MIGRA-ZEN RELIEF PLUS
Dietary Supplement: Placebo for Migrazen relief plus — 2 capsule dose per 24 hours for 90 days
  Arms: Placebo for Migra zen plus

SUMMARY:
The purpose of this study is to study MIGRA-ZEN RELIEF PLUS, an all-natural herbal dietary supplement product, with respect to alleviating and/or stopping migraine headache pain compared to a placebo when used prophylactically. This study will involve subjects suffering from chronic migraine headaches.

DETAILED DESCRIPTION:
The purpose of this 90-day, randomized, double-blind, placebo controlled study is to evaluate the efficacy of an all-natural herbal dietary supplement product, (Investigational Product, or IP), with respect to alleviating and/or stopping migraine headache pain compared to a placebo when used prophylactically every day, and to evaluate the safety/risk of its use by observing the absence/presence of adverse event (AE/SAE) reports and the normalcy of blood work, urinalysis, and liver enzyme tests. The primary end-point is the time-course and depth of the frequency reduction of migraine attacks. The secondary end-points will be the absence/presence of detectable adverse liver function and urinalysis test results as well as the dearth/abundance of AE/SAE reports that may indicate patient safety/risk when using the IP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older.
* Prior to this study subject must have been diagnosed with migraines according to IHS criteria by a qualified healthcare professional with some experience in the diagnosis of migraines and have suffered with them for one year prior to the start of the study.
* Migraine symptoms/attacks must have presented for a minimum of the last consecutive three (3) months at a minimum average frequency of six (6) times per month and must have been severe-extreme (grade 7-10) on a linear scale of 0-10, where 0=no pain and 10=unbearable maximum pain.
* Subjects who are able to follow the protocol as designed by RZN Nutraceuticals, Inc. and Teva Pharmaceutical Industries.
* Generally good health

Exclusion Criteria:

* Subjects currently taking any prophylactic treatment for migraine headaches
* History of head trauma or brain cancer.
* Candidate subjects with any medical condition that, in the opinion of the investigators or intake staff, would jeopardize the safety of the patient, affect the validity of the data collected from the subject, or would challenge the subject's ability to complete the study protocol for 90 days.
* Known renal insufficiency or kidney disease of any grade
* Any illness causing severe coughing so as to avoid introducing "coughing migraine" per IHS classification 4.2, G44.803.
* History of drug addiction.
* Females of child-bearing potential who do not practice medically acceptable methods of contraception surgical, sterilization, intrauterine device (IUD), hormonal preparations or double barrier method (e.g. condom or diaphragm and spermicide)
* Subjects with uncontrolled hypertension (e.g. BP>150/100).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The reduction of migraine attacks | 90 Days
  The time-course and depth of the frequency in the reduction of migraine attacks

SECONDARY OUTCOMES:
AEs SAEs | 90 days
  The secondary end-points will be the absence/presence of detectable adverse liver function and urinalysis test results as well as the dearth/abundance of AE/SAE reports that may indicate patient safety/risk when using the IP.

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Mosek, MD, Principal Investigator — Saurasky Tel Aviv Medical Center, Israel
Locations (2):
- Israel (2):
  - Rabin Medical Centre, Petah Tikva
  - Sourasky Medical Centre, Tel Aviv